CLINICAL TRIAL: NCT04686240
Title: Doppler Ultrasonographic Assessment of Fetal Internal Thoracic Artery Indexes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Yakıştıran, specialist, Ankara City Hospital Bilkent
Other Study IDs: internalthoracicarterydoppler
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Pregnancy Related; Fetal; Circulation
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the feasibility of visualizing the internal thoracic artery (ITA), establishing the normogram for ITA pulsatility index (PI), resistance index (RI) and acceleration/ejection time (AT/ET) at 24-32 weeks.

DETAILED DESCRIPTION:
Background: The internal thoracic artery arises from the subclavian artery as the first branch. It travels downward on the inside of the rib cage and then gives off six main branches; mediastinal, thymic, pericardiacophrenic, sternal, perforating and intercostal branches.

In literature, there are so many articles that have been focused on thymus size in pregnancies complicated with diabetes mellitus, fetal growth restriction, preterm rupture of membranes and so on. To the best of our knowledge, there is no paper about fetal ITA whose branch are feeding vessel of thymus and ITA Doppler velocity. The arteries supplying the thymus are branches of the internal thoracic, and inferior thyroid arteries. As far as it has been known, growing of a tissue depends on increased blood flow. Before detecting possible blood-flow changes in fetuses complicated with great obstetrics patologies, the investigators should obtain normal values of ITA Doppler velocity.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* having no fetal anomalies
* healthy pregnant women age >17 and <45 years
* between 24th-32nd gestational weeks

Exclusion Criteria:

* fetuses with congenital aneuploidy or structural malformation
* underlying chronic diseases
* pregnant women complicated with gestational diabetes, Type 1-2 DM, hypertension (pregnancy-induced; chronic; preeclampsia), malignancy
* pregnancy complicated with preterm premature rupture of membranes, preterm labour, fetal growth restriction and another obstetric complication

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant
Study Population: healthy fetuses between 24th and 32nd gestational weeks
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Doppler indices for internal thoracic artery | Between 24th and 32nd gestational weeks
  Doppler indices (pulsatility index, resistance index, acceleration and ejection time)
assessment of fetal thymus size | Between 24th and 32nd gestational weeks
  volume and perimeter and transvers diameter

CONTACTS AND LOCATIONS:
Overall Officials: betül yakıştıran, MD, Principal Investigator — Ankara City Hospital Bilkent; aykan yücel, professor, Principal Investigator — Ankara City Hospital Bilkent; mihriban alkan, MD, Principal Investigator — Ankara City Hospital Bilkent; seval erdinç, assoc prof, Principal Investigator — ankara city hospitalBilkent